CLINICAL TRIAL: NCT02081352
Title: Phase IV Prospective, Multi-Center, Randomized, Single-Blind, Active and Standard Care-Controlled Study of DermaPure™ in Patients With "Hard to Heal" Chronic, Neuropathic Diabetic Foot Ulcers With Crossover Design for Standard Care Arm
Brief Title: A Comparative Efficacy Study of DermaPure™ to Treat Diabetic Foot Ulcers
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TRx Wound Care Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRG-H01-01
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Diabetic Foot Ulcers
Keywords: Dermis; Diabetic foot ulcers; Skin substitutes; Decellularized
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DermaPure™ (Active Comparator): DermaPure™ in combination with standard care comprising surgical debridement, covered by a non-adherent silicone wound contact layer, a wound cavity filler (if required), a secondary foam wound dressing and appropriate off-loading footwear.
  Interventions: Other: DermaPure™
- Standard care (Sham Comparator): Standard care comprising surgical debridement, covered by a non-adherent silicone wound contact layer, a wound cavity filler (if required), a secondary foam wound dressing and appropriate off-loading footwear.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: DermaPure™ — A minimally manipulated human tissue regulated as "human cells, tissues, and cellular and tissue-based products" (HCT/Ps)
  Arms: DermaPure™
Other: Standard care
  Arms: Standard care

SUMMARY:
This study has been designed to help determine how safe and effective DermaPure™ may be in treating hard-to-heal diabetic foot ulcers compared to the current standard of care.

DETAILED DESCRIPTION:
DermaPure™ is a decellularized dermal skin substitute using the Tissue Regenix dCELL® patented Technology to remove cells and other components from human and animal tissue while maintaining the native structural and biomechanical properties. The primary objective of the study is to establish the wound healing performance and safety of DermaPure™ over a 12 week period, when administered to "hard to heal" chronic, neuropathic diabetic foot ulcers. This study has been designed to compare the performance of DermaPure™ (in combination with standard care) versus standard care alone.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes with HbA1c ≤12%
* Adequate perfusion
* A full thickness chronic, neuropathic diabetic foot plantar ulcer defined by Texas or Wagner classification.
* Target ulcer decreases in size (surface area) by less than 30% in the 2 week screening period.

Exclusion Criteria:

* BMI greater than 45kg/m2.
* Presence of infection
* Presence of necrosis, purulence or sinus tracts that cannot be removed by aggressive debridement.
* A clinical diagnosis of an active/acute Charcot neuroarthropathy. Inactive/chronic Charcot does not exclude the patient.
* Therapy with any investigational agent or drug within 4 weeks preceding the screening visit.
* More than 2 weeks treatment with immunosuppressive agents within 3 months of enrollment.
* Evidence of malnutrition as confirmed by serum pre-albumin level at screening.
* Evidence of drug or alcohol abuse,

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-11 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of wound closure | 12 weeks
  The incidence of full wound closure at or before 12 weeks, where full wound closure is defined as "100% re-epithelialization, without drainage, that has been confirmed at two study visits up to 14 days apart".

SECONDARY OUTCOMES:
Rate of wound healing | 12 weeks
  Percentage reduction in ulcer area and volume, weekly up to Week 12 compared to baseline.
Quality of wound healing | 4 weeks
  Cellular profile through histological analysis of wound biopsies at Week 4 compared to baseline

OTHER OUTCOMES:
Rate of wound healing in crossover arm | 6 weeks
  Percentage reduction in ulcer area and volume, weekly up to Week 18 compared to Week 12 for a subset of subjects who receive first application of DermaPure™ at Week 12 (Crossover arm).

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Carl T. Hayden Medical Research Foundation, Phoenix, Arizona
  - Associated Foot & Ankle Specialists, Phoenix, Arizona
  - University of Miami Hospital, Miami, Florida
  - NYU Langone Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Futuro Clinical Trials, LLC, McAllen, Texas